CLINICAL TRIAL: NCT05660694
Title: Comparison of Triamcinolone With Pentoxifylline and Vitamin- E Efficacy in the Treatment of Stage 2 and 3 Oral Submucous Fibrosis: A Clinical Trial
Brief Title: Comparison of Triamcinolone With Pentoxifylline and Vitamin- E Efficacy in the Treatment of Stage 2 and 3 Oral Submucous Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Abhishek Lal, Dr. Abhishek Lal, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Treatment of OSF stage 2 and 3
Record Dates: First submitted 2022-12-04; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Triamcinolone; Pentoxifylline; Vitamin E; Oral Submucosa Fibrosis; Tumor
MeSH Terms: conditions — Neoplasms | interventions — Triamcinolone; Pentoxifylline; Vitamin E

STUDY DESIGN:
Intervention Model Description: Group 1: Triamcinolone Group 2: Pentoxifylline
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Triamcinolone (Experimental): Injection steroid Triamcinolone 400mg with lidocaine 1:1 was given twice a week for 4 weeks in bi-lateral buccal mucosa in multiple sites
  Interventions: Drug: Triamcinolone
- Group 2: Pentoxifylline with Vitamin E (Experimental): Pentoxifylline 40mg twice a day along with vitamin E supplement one tablet per day for 4 weeks
  Interventions: Drug: Pentoxifylline with Vitamin E

INTERVENTIONS:
Drug: Triamcinolone — Comparison of Triamcinolone with Pentoxifylline and Vitamin- E Efficacy
  Arms: Group 1: Triamcinolone
Drug: Pentoxifylline with Vitamin E — Comparison of Triamcinolone with Pentoxifylline and Vitamin- E Efficacy
  Arms: Group 2: Pentoxifylline with Vitamin E

SUMMARY:
To compare the efficacy of Triamcinolone with Pentoxifylline and Vitamin E in patients with stage two and three oral submucous fibrosis.

DETAILED DESCRIPTION:
To compare the efficacy of Triamcinolone with Pentoxifylline and Vitamin E in patients with stage two and three oral submucous fibrosis.

It was a randomized control clinical trial to compare efficacy of injection steroids versus pentoxifylline and vitamin E in the treatment of stage 2 and 3 OSF patient. Total 40 patients who presented with signs and symptoms of OSF were enrolled in our study that was evaluated over the period of (January 2020 to September 2021). Parameters taken in the study were age and mouth opening. Descriptive statistics and paired t-test were used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically diagnosed OSMF who have not undergone any treatment of OSMF in past
* Patients willing to quit their tobacco chewing habit, gutkha areca nut smoking
* Patients who are ready to attend regular follow-ups

Exclusion Criteria:

* Patients who have undergone any treatment for OSF in past
* Patients with any evidence of cardiac, gastrointestinal, kidney, metabolic disorders, pregnant and lactating women's
* Patients with any co-existing disorder of the orofacial region other than OSF which may interfere with the study protocol

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Group 1: Triamcinolone measuring mouth opening using calibrated Vernier Caliper | 21 months
  Measuring mouth opening measuring mouth opening using calibrated Vernier Caliper by recording in millimeters the maximum mouth opening
Group 2: Pentoxifylline with Vitamin E measuring mouth opening using calibrated Vernier Caliper | 21 months
  Measuring mouth opening measuring mouth opening using calibrated Vernier Caliper by recording in millimeters the maximum mouth opening

CONTACTS AND LOCATIONS:
Locations (1):
- Altamash Institute of Dental Medicine, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided